CLINICAL TRIAL: NCT01627080
Title: Cardiac Biomarker Study in Esophageal Cancer Patients Treated With Chemotherapy and Radiation
Status: Withdrawn | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-0004
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Esophageal Cancer
Keywords: Esophagus; Esophageal Cancer; Radiation therapy; RT; Chemotherapy; Mid thoracic tumor; Distal esophageal tumor; Gastroesophageal junction tumor; Cardiac biomarkers
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draws include troponin I, NT-proBNP, and BNP.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Biomarkers: Patients with histologically proven esophageal cancer to be treated with radiation therapy with concurrent chemotherapy to a final dose of >/=40 Gy included in this study at UT MD Anderson Cancer Center in Houston, Texas.
  Interventions: Other: Cardiac Biomarker Blood Draws

INTERVENTIONS:
Other: Cardiac Biomarker Blood Draws — Blood (about 1 teaspoon) drawn to measure cardiac biomarkers at the following time points: within 12-24 hours of the start of radiation, one (1) time during the third week of radiation, within 48 hours after completion of radiation, and about 1 to 2 months after completion of radiation therapy.

SUMMARY:
The goal of this clinical research study is to learn if the radiation that you will receive for esophageal cancer may cause the heart to create more proteins called cardiac biomarkers.

When cardiac biomarkers are above normal levels, there may be heart damage. The relationship between cardiac biomarkers and radiation therapy has not been well studied. Learning more about this relationship may lead to better ways to check the heart during radiation therapy and predict heart problems.

DETAILED DESCRIPTION:
If you are found to be eligible and you agree to take part in this study, you will have baseline tests. The following tests and procedures will be performed within 1-2 weeks from the start of radiation:

* You will be asked about any other health problems you may have.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn to measure cardiac biomarkers.
* You will have an electrocardiogram (ECG) to check your heart function.
* If the study doctor thinks it is needed, you will have an exam by a cardiologist (a doctor who diagnoses and treats heart problems) who will check the results of your ECG.

Study Visits:

Blood (about 1 teaspoon) will be drawn to measure cardiac biomarkers at the following time points:

* Within 12-24 hours of the start of radiation
* One (1) time during the third week of radiation
* Within 48 hours after completion of radiation

Follow-Up:

About 1 to 2 months after you complete radiation therapy, depending on when you and your doctor decide, you will return to the clinic. The following tests and procedures will be performed:

* Blood (about 1 teaspoon) will be drawn to measure cardiac biomarkers.
* You will have an ECG.

Length of Study Participation:

You will be off study after your follow-up visit.

You will no longer be able to take part in the study if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

This is an investigational study. Using cardiac biomarkers to check the heart during radiation therapy to predict future heart problems is considered investigational.

Up to 100 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven esophageal cancer to be treated with RT with concurrent chemotherapy to a final dose of >/=40 Gy will be included in this study.
2. Patients with mid thoracic, distal esophageal, and gastroesophageal junction tumors.
3. All patients must sign a study-specific informed consent form. If the patient's mental status precludes his/her giving informed consent, written informed consent may be given by the patient's legal representative.
4. Age >/= 18
5. Women of childbearing potential (A woman of child-bearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months [i.e., who has had menses at any time in the preceding 24 consecutive months]. For women of childbearing potential, a blood pregnancy test must be performed within 72 hours prior to the start of protocol treatment.
6. Induction chemotherapy allowed.
7. Being able to meet radiation dose constraints of at-risk organs.

Exclusion Criteria:

1. Patients who receive cardiotoxic drugs, such as trastuzumab or adriamycin as part of their chemotherapy regimen.
2. Patients with recent myocardial infarction in the past month, decompensated heart failure or myocarditis/pericarditis in the past month.
3. Patients with renal failure indicated by a glomerular filtration rate (GFR) < 30 mL/min/1.73sq.m.
4. Patients in the intensive care unit (ICU).
5. Patients with systemic sepsis.
6. Patients with acute pulmonary embolism in the past month.
7. Women who are pregnant or nursing are not eligible as treatment involves unforeseeable risks to the fetus or child.
8. Inability to obtain histologic proof of malignancy.
9. Patients with proximal / cervical esophageal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven esophageal cancer to be treated with radiation therapy with concurrent chemotherapy to a final dose of >/=40 Gy included in this study at UT MD Anderson Cancer Center in Houston, Texas.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Cardiac Biomarker Elevation with Radiation Therapy | Within 24 hours after first fraction of radiation therapy (RT), during 3rd week of RT (fraction 11-15), within 48 hours of RT completion (fraction 26-28).
  Descriptive statistics used to summarize change from baseline in enzyme levels at each time point (beyond baseline). Each enzyme examined separately. Pearson or Spearman correlation coefficient used to examine correlation between changes in cardiac biomarkers from baseline in enzyme level at each time point and mean radiotherapy dose or cumulative dose to heart. Linear mixed effects regression model used to model longitudinal change in cardiac biomarker from baseline as a function of cumulative radiation to the heart, radiation modality (Protons vs Photons), and time.

SECONDARY OUTCOMES:
Incidence of Adverse Cardiac Outcomes | Within 24 hours after first fraction of radiation therapy (RT), during 3rd week of RT (fraction 11-15), within 48 hours of RT completion (fraction 26-28).
  Incidence of adverse cardiac outcomes tabulated including myocardial infarction, heart failure, arrhythmias, all-cause and cardiac-specific mortality at same time points used to analyze cardiac biomarker levels.

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Lin, MD,PHD, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org